CLINICAL TRIAL: NCT06464458
Title: Optimizing the Management of Sickle Cell Patients on Hydroxyurea: The Value of Therapeutic Pharmacological Monitoring
Acronym: OPTIMDREP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8100
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell; Hydroxyurea; Therapeutic drug monitoring; Pharmacokinetics; SIKLOS®; HYDREA®
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Pharmacokinetics results of patients in Arm A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control) (No Intervention): DDepending on haematological tolerance (MTD), dose adjustment is proposed if necessary to achieve neutrophils between 1.5 - 3.0 G/L and reticulocytes between 100 - 200 G/L, without exceeding the maximum dose of 35 mg/kg. The titration step is 5 mg/kg except in the case of CrCl ≤ 60 ml/min; 2.5 mg/kg step in this case.
- Arm B (Experimental): HU dose adaptation according:
  * HU AUC with a target AUC and subject to haematological tolerance.
  * T2H (at V2, V3, V4), subject to haematological tolerance.
  Interventions: Other: management on hydroxyurea by therapeutic pharmacological monitoring

INTERVENTIONS:
Other: management on hydroxyurea by therapeutic pharmacological monitoring — HU dose adaptation according:
  * HU AUC with a target AUC and subject to haematological tolerance.
  * T2H (at V2, V3, V4), subject to haematological tolerance.
  Arms: Arm B

SUMMARY:
Brief Summary: * A short description of the clinical study, including a brief statement of the clinical study's hypothesis, written in language intended for the lay public.

Limit: 5000 characters.

Severe forms of sickle cell syndrome are characterized by the occurrence of repeated vaso-occlusive crises (CVO), early complications and a high morbidity and mortality in these patients. Intensified management is then required, with the introduction of hydroxyurea treatment and then, if it proves ineffective, a transfusion program or even a haematopoietic stem cell allograft. These latter treatments present significant risks of adverse effects for the patient (haemochromatosis, erythrocyte alloimmunisation for the transfusion program, risk of GVH, chemotherapy-related toxicity, MVO for the allograft).

Hydroxyurea (HU) is the first treatment based on the specific pathophysiology of sickle cell disease. It is the first line of therapeutic intensification for adult patients and children (age ≥ 2 years) with major sickle cell disease. By mainly increasing the percentage of fetal haemoglobin (HbF), HU decreases the frequency of CVO, complications, hospitalizations and prolongs the life expectancy of patients.

The initial dose of HU, recommended by the ANSM, is 15 mg/kg/d once daily. However, the optimal dose cannot be predicted at the start of treatment, which is why a dosage adjustment is essential. The usual dose is between 15 and 35 mg/kg per day.

Typically, the dose is increased every 3 months until a mild myelosuppression tolerated by the patient is reached, indicating that the maximum tolerated dose (MTD) has been reached. When the dose of HU has reached the MTD, the ratio of clinical (reduced frequency of vaso-occlusive attacks) and biological (better % of HbF) benefits to risk (toxicity) is optimal for the patient.

The disadvantages of this practice are that:

* dose escalation can be long (9-12 months)
* clinicians may be reluctant to escalate HU to MTD
* patients are treated sub-optimally during the therapeutic adaptation period.

Recent work has shown that it is beneficial for the patient to adjust the initial dose using a pharmacological therapeutic approach in addition to monitoring haematological tolerance.

Thus, by customizing the dose of HU using an area under the curve (AUC) measurement at the initial intake of HU at a standardized dose (20 mg/kg/day), the MTD would be achieved in a faster time frame of 6-9 months.

The primary objective of our trial is to identify the methodology that will most effectively decrease the time to reach the MTD (therapeutic target). The immediate benefit will be a reduction in CVO which is the major clinical problem and leads to a risk of complications in sickle cell disease.

DETAILED DESCRIPTION:
• Information visit (V0 - 7 days to V0 - 6 months) Patients seen in a routine consultation will be informed about the project in an interview with the doctor, and the information leaflet will be given to the patient and/or his/her parents. In case a patient is admitted to a conventional ward, information about the study will be given in a meeting with the doctor. They will have 7 days to think about it. If they agree to participate in the study, a second appointment will be made, with sufficient time for reflection, for the signing of the consent form.

The information and consent of minor patients will be the subject of an adapted procedure. In example, a specific notice will be provided for children of a comprehensible age (under 11 years). In addition, an information leaflet will be provided and adapted to the level of understanding of each age category for minor patients (11 to 16 years; adults).

• Inclusion visit (V0 - 7 days to V0 - 173 days) Prior to any research-related examination, the free, informed and signed consent of the parent(s) and the minor, if applicable, the legal representative or the patient if of age, is obtained after a reflection period has been respected.

The date on which the subject (or the parent(s) and the minor, if applicable, or the legal representative) agreed to participate in the research is noted in the medical file, as is the date of any objection to participation, if applicable.

In addition, the consent of the minor subject will be sought if he/she reaches his/her majority during his/her participation in the research.

During this visit, the eligibility criteria will be checked and if the patient is eligible, he/she and/or his/her legal representatives will be able to sign the consent.

- Randomisation visit (V0 visit)

The following examinations/actions will be performed to confirm the subject's eligibility for further participation in the study:

* Collection of medical, surgical and lifestyle history
* Physical examination (weight, height, blood pressure, heart rate, medical examination)
* Randomisation is then carried out by the investigator (or a delegated person) via the Internet, using the Cleanweb platform, which is accessed by the investigator or the delegated person using their personal access codes. It allows the allocation of the treatment group, i.e.:

  * Arm A (Control): Dose adjustment based on haematological assessment
  * Arm B (Experimental): Dosage adjustment based on AUC at D1, then control of the pharmacokinetic target by T2H and monitoring of haematological tolerance.
* HU is then taken orally:

The drug should be taken under the usual conditions for children:

Samples are then taken on EDTA tubes They will allow the calculation of the patient's exposure to the drug (AUC).

The patient is given a prescription for a test to be carried out in the city at D15 after the introduction of the HU or after the dosage has been adjusted, in order to assess tolerance (MTD).

• Visit V1 (M3) As at the first visit, the usual clinical and biological examinations are performed.

The results of the PK assay and tolerance (MTD) being available, a dosage adjustment is proposed according to the patient's randomisation arm and without exceeding the maximum dose of 35 mg/kg:

* Arm A: adjustment in 5 mg/kg steps (or 2.5 mg/kg if CrCl<60ml/min) according to maximal toxic dose (MTD).
* Arm B: Adaptation according to V1 HU AUC. A prescription for a CBC to be carried out in the city at D15 after the dosage adjustment is given to the patient in order to assess tolerance.

  * V2 visits (M6 +/- 1 month) As at the first visit, the usual clinical and biological examinations are performed.

The results of the PK assay and tolerance (MTD) being available, a dosage adjustment is proposed according to the patient's randomisation arm and without exceeding the maximum dose of 35 mg/kg:

* Arm A: adjustment in 5 mg/kg steps (or 2.5 mg/kg if CrCl<60ml/min) according to maximal toxic dose (MTD).
* Arm B: Adaptation according to V1 HU AUC. A prescription for a CBC to be carried out in the city at D15 after the dosage adjustment is given to the patient in order to assess tolerance.

  * Visit 3 (M9 +/- 1 month) and visit 4 (M12 +/- 1 month):

As at the first visit, the usual clinical and biological examinations are performed.

The results of the PK assay and tolerance (MTD) being available, a dosage adjustment is proposed according to the patient's randomisation arm and without exceeding the maximum dose of 35 mg/kg:

* Arm A: adjustment in 5 mg/kg steps (or 2.5 mg/kg if CrCl<60ml/min) according to maximal toxic dose (MTD).
* Arm B: Adaptation according to V1 HU AUC. A prescription for a CBC to be carried out in the city at D15 after the dosage adjustment is given to the patient in order to assess tolerance.

  • Visit V5 (M15) On the day of visit 5, the patient is welcomed in the department.
* HU is taken at the usual dosage.
* Then the pharmacokinetic samples are taken.

Subsequent follow-up:

The study does not require specific follow-up. However, patients will continue to be followed by their referring physician in a day hospital or in a consultation every 3 months, according to the usual management modalities.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged between 2 and 35 years.
* For very young children hydroxyurea is only initiated in cases of severe sickle cell disease.
* Sickle cell genotype: HbSS
* Subjects who have been hospitalised for CVO in the last 3 months and for whom HU treatment is to be initiated and/or whose treatment is not balanced or is less than 30 mg/kg, regardless of the length of treatment
* For a woman of childbearing potential:
* Negative blood pregnancy test at the inclusion visit
* Patient accepting highly effective contraception for the duration of study participation and 182 days after discontinuation of the study or treatment.
* Initiation of HU treatment in a patient requiring intensification of therapy in the context of sickle cell disease
* Patient hospitalised (e.g. vaso-occlusive crisis) and/or whose HU treatment is not balanced (MTD not reached)
* Informed consent signed, as appropriate, by :

  * The patient and/or
  * The holder(s) of parental authority and the minor subject if capable of discernment
* Subject affiliated to a social health insurance scheme or beneficiary
* Subject who has been informed of the results of the prior medical examination, and/or of whom the holder(s) of parental authority has (have) been informed
* Subject able to understand the objectives and risks of the research and to give dated and signed informed consent

Exclusion criteria:

* HU patient who has achieved MTD (based on haematological criteria) or is not therapeutically ineffective or hydroxyurea dosage > 35 mg/kg/day.
* Refusal to accept the use of a highly effective contraceptive method as defined during HU treatment and for 182 days for females and 92 days for males following such treatment (fertile patients only)
* Patient with a parental plan within 18 months
* Hypersensitivity to the active substance or to any of the excipients of the medicinal product
* Severe hepatic impairment
* Severe renal insufficiency
* Toxic signs of myelosuppression
* Neutrophils < 1500/mm3
* Platelets < 80 000/mm3
* Haemoglobin < 4.5 g/dL
* Reticulocytes < 80,000/mm3 if haemoglobin concentration < 9 g/dL
* Patient with transfusion, exchange transfusion or erythropoietin administration within 3 months of inclusion
* Patient with HIV
* Unable to give subject informed information (subject in emergency situation)
* Inability of the subject to undergo the medical follow-up of the trial for geographical, social or psychological reasons
* Subject under guardianship or curatorship
* Pregnancy or breastfeeding in the case of adolescents or adults
* Subject in an exclusion period (determined by a previous or ongoing study)
* Concurrent inclusion in another drug study
* Subject under court protection

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the time to obtained MTD in 2 groups of sickle cell patients on hydroxyurea with different treatment follow-up methodology: MTD follow up or therapeutic pharmacological monitoring | Theoretical start date: January 2023 Duration of inclusion period: 30 months Duration of participation of each subject: 16 months Total study duration: 46 months
  - Arm A (Control): The dosage adjustment is quarterly from M3 onwards and will be made on hematological (WBC) tolerance. The increase of the dosage in HU will be 5 mg/kg every 3 months (or 2.5 mg/kg in case of renal insufficiency with ClCr ≤ 60 ml /min) until MTD is achieved and within a limit of 35 mg/kg/day (max 2500mg).
  - Arm B (Experimental): Dose adjustment will be done at the M3 visit based on the results of the Pharmacokinetic analysis (AUC) performed on the day of the first HU intake after inclusion. At the quarterly visits V1 (3 months) to V4 (12 months), a HU assay at time T = 2H associated with monitoring of hematological monitoring of hematological tolerance will be performed to verify the pharmacokinetic stability in the child after the dosage adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Paillard, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Strasbourg University Hospital, Strasbourg, France